CLINICAL TRIAL: NCT00182858
Title: Tissue Procurement for Biomedical Research
Status: Recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903322; 03-AG-N322; NCT01927796 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-09-29

CONDITIONS: Normal Volunteers
Keywords: Biologic Sample Collection; Tissue Procurement; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants will be 18 years or older that are Healthy Volunteers or have been identified by the investigator and/or physician to have a condition of interest for exploratory studies related to the participant s illness or other feature that offers the possibility of creating information that leads to scientifically useful and important studies.

SUMMARY:
The need to obtain human tissue for methods development and disease correlation is frequent in Biomedical Research Center laboratories. This protocol is designed to create the opportunity to obtain such tissue samples including: blood, urine, saliva, sweat, feces, hair and nail clippings, nasal scraping, muscle, fat, skin and taste buds. It may also include samples taken during a surgical procedure, including: fluid from around the spinal column, heart, lungs and abdomen; fat, muscle, connective tissue and organs (liver, bladder, heart, kidney and skin).

Information derived from such studies is for research purposes only and is not provided to the participants or their health care provider. Samples will be coded (no names) and identifying information linking the participant to the sample will be maintained in a secure location by the P.I. and Study Coordinator.

Participants will be 18 years or older and have been identified by the investigator and/or physician to have a condition of interest for exploratory studies related to the participant s illness or other feature that offers the possibility of creating information that leads to scientifically useful and important studies. Participants could also be healthy volunteers, willing to provide their samples. These samples could be requested by an investigator to be used as age, gender, race and/or ethnicity-matched controls or to calibrate or compare and contrast across lab equipment. Participants will be excluded if obtaining the sample would be over and above usual clinical care, would result in excessive blood loss, or the individual is unable to provide informed consent.

The expected outcome is to provide investigators with the opportunity to obtain tissues of interest for laboratory evaluation....

DETAILED DESCRIPTION:
The need to obtain human tissue for methods development and disease correlation is frequent in Biomedical Research Center laboratories. This protocol is designed to create the opportunity to obtain such tissue samples including: blood, urine, saliva, sweat, feces, hair and nail clippings, nasal scraping, muscle, fat, skin and taste buds. It may also include samples taken during a surgical procedure, including: fluid from around the spinal column, heart, lungs and abdomen; fat, muscle, connective tissue and organs (liver, bladder, heart, kidney and skin).

Information derived from such studies is for research purposes only and is not provided to the participants or their health care provider. Samples will be coded (no names) and identifying information linking the participant to the sample will be maintained in a secure location by the P.I. and Study Coordinator.

Participants will be 18 years or older and have been identified by the investigator and/or physician to have a condition of interest for exploratory studies related to the participant s illness or other feature that offers the possibility of creating information that leads to scientifically useful and important studies. Participants could also be healthy volunteers, willing to provide their samples. These samples could be requested by an investigator to be used as age, gender, race and/or ethnicity-matched controls or to calibrate or compare and contrast across lab equipment. Participants will be excluded if obtaining the sample, would result in excessive blood loss, or the individual is unable to provide informed consent.

The expected outcome is to provide investigators with the opportunity to obtain tissues of interest for laboratory evaluation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 or older.
* Identified by the investigator , researcher, or physician to have a condition of interest for exploratory studies related to the participant s illness or other feature that offers the possibility of generation of hypotheses for future study.
* Healthy volunteers, willing to provide their samples.

EXCLUSION CRITERIA:

* The participant would be subjected to diagnostic and/or therapeutic procedures that are not necessary for clinical management.
* Excessive blood loss if this phlebotomy plus other research participation and/or clinical evaluation will result in blood loss of greater than 1 unit (400 ml, 1 pint) over an 8-week period.
* Inability to give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any healthy volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2003-06-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31

PRIMARY OUTCOMES:
Provide the investigators the opportunity to obtain tissues for laboratory evaluation with the goal of either better understanding a disease or design a scientific study to better understand or treat a disease. | Ongoing
  The goal is to assist in either the better understanding of a disease or to design a scientific study to better understand or treat a disease.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The NIA IRP is discussing the plan to make IPD available. A final decision has not been made.